CLINICAL TRIAL: NCT00222014
Title: TIPS (With Coated Stents) OR PARACENTESIS + ALBUMIN ADMINISTRATION FOR THE TREATMENT OF REFRACTORY ASCITES IN PATIENTS WITH CIRRHOSIS : A RANDOMIZED TRIAL COMPARING SURVIVAL, QUALITY OF LIFE AND NUTRITIONAL STATUS
Brief Title: TIPS With Coated Stents for Refractory Ascites in Patients With Cirrhosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Ministry of Health, France (Other Government); GORE Laboratory (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0402308; PHRC
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Cirrhosis
Keywords: Refractory ascites; Cirrhosis; Paracentesesis
MeSH Terms: conditions — Fibrosis; Ascites | interventions — Portasystemic Shunt, Transjugular Intrahepatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): TIPS réalisé avec prothèse couverte de PTFE
  Interventions: Procedure: TIPS
- 2 (Active Comparator): Paracenthese and albumine perfusion
  Interventions: Procedure: Paracenthese

INTERVENTIONS:
Procedure: TIPS — Transjugular intrahepatic portosystemic shunt with covered PTFE
  Arms: 1
Procedure: Paracenthese — Paracenthese
  Arms: 2

SUMMARY:
The main end point of the study is to assess survival in cirrhotic patients with refractory ascites treated by TIPS (using PTFE covered stents) vs patients treated by paracentesis + albumin infusion.

DETAILED DESCRIPTION:
Diagnostic evaluation before randomisation includes assessment of clinical hepatic encephalopathy, usual blood tests, and Doppler-ultrasonography of the abdomen. Inclusion and exclusion criteria will be checked during the inclusion visit. Informations concerning the trial will also be given. After the investigator receives written informed consent, randomisation will be performed online. Randomisation will be centralized, equilibrated for each center, stratified according to whether cirrhosis is alcoholic or not and adjusted every ten patients.

I Treatments

1. TIPS :

   TIPS will be performed under sedation or general anesthesia with tracheal intubation according to the usual policy of participating centers. Pre-tips portosystemic pressure gradient and diameter of the shunt must be notified.

   However, for homogeneity reasons the following will be adhered:

   A 10 mm Viator stent will be used, that will be dilated to 8 or 10 mm according to the hemodynamic response. The aim will be to reduce portal pressure gradient (PPG) below 12 mmHg. Ideal PPG should be 7-8 mmHg.
2. Paracentesis + albumin infusion :

After a paracentesis > 3 liters, 8 g of Albumin per liter of extracted ascites must be infused.

If possible, analysis of ascitic fluid will be performed after each paracentesis for biochemical, cytological and bacterial analyses.

II Follow up

1. In all patients:

   Low salt diet (2 - 4 g/j). Follow up of the patient is as usual. Patients will have a clinical examination at 1 month and then every 3 months up to 1 year. At each visit, clinical and biochemical variables needed to calculate Child-Pugh score will be recorded.

   Doppler ultrasonography will be performed at the beginning, 6 and 12 months. Patients will be followed 1 year or until liver transplantation or death.
   1. Nutritional status evaluation:

      * Weight: M0, M3, M6, M9, M12
      * Anthropometrics measurements: M0, M3, M6, M12: they will include : triceps skinfold thickness, biceps skinfold thickness, brachial circumference.
      * Biochemical parameters: M0, M3, M6, M12: they will include : albumin, pre-albumin, orosomucoïde, C-reactive protein, haptoglobin, natriuresis, 24 hour urinary excretion of creatinine. Four blood samples will be collected and conserved for a posteriori analysis if required (transferrin, retinol binding protein, leptin, hormonal dosages). These analyses will be centralized in Toulouse (Toulouse center will be charged for the shipment of those blood samples).
      * Physical parameters: dual energy x-ray absorptiometry M0, M12
      * Grip test M0, M6, M12 [16, 17].
   2. Quality of Life :

   SF-36 (Short Form 36 (SF-36) Health Survey Questionnaire) at inclusion and then every three months [18, 19].
2. Paracentesis + albumin infusion group:

   Patients included in this group will be treated by paracentesis whenever required. Eight grams of albumin per liter of ascites extracted will be infused when more than 3 liters of ascitic fluid will be removed.
3. TIPS group :

When shunt dysfunction will be suspected because of relapse of ascites or incomplete response 2 months after the procedure, an angiography and PPG measurement will be performed. If shunt dysfunction is confirmed, angioplasty or PTFE re-stenting will aim at reducing PPG below 12 mmHg.

III Definition of treatment failure:

After TIPS: relapse of ascites requiring at least 2 paracenteses or persistence after 2 months will be considered as treatment failure. A hemodynamic and angiographic control will be performed. Patients will be treated by refection of the shunt. If severe encephalopathy occurs and persists despite treatment, the diameter of the shunt should be decreased or the TIPS occluded. Total occlusion of the shunt or relapse of ascites after the reduction of its diameter will be also considered treatment failures.

In the group treated by paracentesis + albumin infusion, patients having more than 6 paracenteses within 3 months will be considered for alternative treatment (TIPS, transplantation). Technical impossibility or refusal of the patient to proceed with paracenteses will be also considered treatment failure. In these cases, a TIPS could also be proposed.

All these patients with treatment failure must be followed up to one year after inclusion

ELIGIBILITY:
Inclusion Criteria:

* patients of both sexes, with cirrhosis, as documented by previous liver-biopsy or usual clinical and biochemical stigmata
* with refractory or recurrent ascites as defined in chapter IV
* who signed the informed consent form

Exclusion Criteria:

* patients not fulfilling inclusion criteria
* patients having needed more than 6 paracenteses within the last 3 months
* patients expected to be transplanted within the next 6 months
* usual contra-indication for TIPS : congestive heart failure NYHA>III or medical history of pulmonary hypertension, portal vein thrombosis, hepatic polycystosis, intra-hepatic bile ducts dilatation, spontaneous clinical recurrent hepatic encephalopathy
* hepatocarcinoma on the expected tract of the shunt
* severe liver failure as defined by : Prothrombin index < 35 % or total bilirubin > 100 micromol/l or Child Pugh Score >12
* serum creatinine > 250 micromol/l
* uncontrolled sepsis
* known allergy to albumin
* pregnant or breast feeding women
* refusal to participate or patient unable to receive informations or to sign written informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2005-05; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Survival at one year | one year

SECONDARY OUTCOMES:
Quality of life, nutritional status, occurrence of complications (other than ascites) secondary to portal hypertension. | one year

CONTACTS AND LOCATIONS:
Overall Officials: BUREAU Christophe, MD, Principal Investigator — University Hospital, Toulouse, France
Locations (4):
- France (4):
  - University Hospital, Angers
  - University Hospital, Lille
  - Hôpital de la Pitié-Salpétrière, Paris
  - Service d'Hépato-Gastro-Entérologie, Hôpital Purpan, Toulouse

REFERENCES:
- [Background] Bureau C, Garcia-Pagan JC, Otal P, Pomier-Layrargues G, Chabbert V, Cortez C, Perreault P, Peron JM, Abraldes JG, Bouchard L, Bilbao JI, Bosch J, Rousseau H, Vinel JP. Improved clinical outcome using polytetrafluoroethylene-coated stents for TIPS: results of a randomized study. Gastroenterology. 2004 Feb;126(2):469-75. doi: 10.1053/j.gastro.2003.11.016. PMID 14762784
- [Derived] Gonzalez-Garay AG, Serralde-Zuniga AE, Velasco Hidalgo L, Flores Garcia NC, Aguirre-Salgado MI. Transjugular intrahepatic portosystemic shunts for adults with hepatorenal syndrome. Cochrane Database Syst Rev. 2024 Jan 18;1(1):CD011039. doi: 10.1002/14651858.CD011039.pub2. PMID 38235907
- [Derived] Bureau C, Thabut D, Oberti F, Dharancy S, Carbonell N, Bouvier A, Mathurin P, Otal P, Cabarrou P, Peron JM, Vinel JP. Transjugular Intrahepatic Portosystemic Shunts With Covered Stents Increase Transplant-Free Survival of Patients With Cirrhosis and Recurrent Ascites. Gastroenterology. 2017 Jan;152(1):157-163. doi: 10.1053/j.gastro.2016.09.016. Epub 2016 Sep 20. PMID 27663604